CLINICAL TRIAL: NCT01256242
Title: A Single Blinded, Multi-center, Randomized, Controlled, Pilot Study to Evaluate the Safety and Performance of Augment™ Rotator Cuff for Primary Surgical Treatment of Full Thickness Rotator Cuff Tears
Brief Title: Pilot Study of Augment Rotator Cuff for Surgical Treatment of Full Thickness Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioMimetic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMTI-2010-03
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: tendon; shoulder; rotator cuff; Glenohumeral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Standard Suture Repair + Augment Rotator Cuff
  Interventions: Device: Augment Rotator Cuff
- Group 2 (Active Comparator): Standard Suture Repair
  Interventions: Procedure: Standard Suture Repair

INTERVENTIONS:
Device: Augment Rotator Cuff — rhPDGF-BB and bovine collagen matrix
  Arms: Group 1
Procedure: Standard Suture Repair — standard suture repair
  Arms: Group 2

SUMMARY:
Study Purpose: To evaluate the safety and performance of Augment Rotator Cuff as a primary surgical treatment for full thickness rotator cuff tears. The hypothesis is that Augment Rotator Cuff will be easy to deliver as an inter-positional graft placed between the rotator cuff tendon and the humeral head providing further enhanced tendon to bone healing without adding any additional safety risk to the patient.

Study Rationale: To evaluate the safety and performance Augment™ Rotator Cuff in surgical intervention of a torn rotator cuff and to obtain preliminary data to support the rationale for a subsequent pivotal clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a repairable rotator cuff tear with an estimated full thickness size of ≥ 2 cm to < 5 cm confirmed with diagnostic MRI in AP or ML dimension
* The subject is independent, ambulatory, and can comply with all post-operative evaluations and visits
* The subject is at least twenty one (21) years of age and considered to be skeletally mature.

Exclusion Criteria:

* The subject has undergone previous rotator cuff repair surgery to the affected shoulder
* The subject has a partial thickness rotator cuff tear
* The subject requires a concomitant subscapularis repair
* The subject requires a concomitant labral repair
* The subject has an irreparable rotator cuff tear
* The subject has an allergy to yeast-derived products or a known bovine collagen allergy
* The subject has implanted metallic devices (cardiac pacemakers, insulin pumps, and nerve stimulators), medically implanted clips or other electronically, magnetically or mechanically activated implants that would contraindicate undergoing an MRI scan of the shoulder
* The subject has tested positive or has been treated for a malignancy in the past or is suspected of having a malignancy or is currently undergoing radiation or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed Augment Rotator Cuff implantation site
* The subject's condition represents a worker's compensation case
* The subject is currently involved in a health-related litigation procedure
* The subject is pregnant or able to become pregnant but not practicing a medically-accepted form of birth control, and/or intending to become pregnant during this study period

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2012-11-16 (Actual); Study Completion 2012-11-16 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | 24 weeks
  The scans were evaluated for degree of re-tears (no re-tears, partial or complete re-tear) by an independent radiologist to assess device integrity and surgical treatment of the rotator cuff tear.
Disabilities of the Arm, Shoulder and Hand (DASH) | 24 weeks
  a self-report questionnaire evaluates the subjects' symptoms and ability to perform activities of daily living, athletic activities and homemaking/work activities. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100
Western Ontario Rotator Cuff Index (WORC) | 24 weeks
  a self-report questionnaire specifically designed to evaluate disability in persons with pathology of the rotator cuff. Each question uses a visual analogue scale (VAS) - which is a straight line, representing a 100-point scale, ranging from 0-100, with a higher score representing lower quality of life.
Constant-Murley Shoulder Outcome Score (CSS) | 24 weeks
  to assess the shoulder and determine at minimum the range of motion (ROM), external rotation and internal rotation, and power score. The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Litchfield, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (4):
- Canada (4):
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario
  - Hand and Upper Limb Clinic - St. Joseph's Health Care London, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - St. Michaels Hospital, Toronto, Ontario

REFERENCES:
- See also: American Academy of Orthopaedic Surgeons — http://www.aaos.org